CLINICAL TRIAL: NCT06178939
Title: Effects of Cognitive Intervention Therapy on Postoperative Delirium in Elderly Non-cardiac Surgical Patients
Brief Title: Effects of Cognitive Intervention Therapy on Postoperative Delirium
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 4-2023-0872
Record Dates: First submitted 2023-12-15; First posted 2023-12-21 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Spinal Stenosis; Disc Herniation; Lung Neoplasms; Carcinoma, Hepatocellular
MeSH Terms: conditions — Spinal Stenosis; Intervertebral Disc Displacement; Lung Neoplasms; Carcinoma, Hepatocellular | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator): The entire process is carried out according to Severance Hospital surgical protocols. The patients of control group will receive education from the research team about the importance of nutrition and exercise before and after surgery.
  Interventions: Procedure: control group
- intervention group (Experimental): For the intervention group, the entire process is carried out according to the Severance Hospital surgical protocol, and the research team provides education before surgery on the importance of nutrition and exercise before and after surgery. In addition, the cognitive training program developed by Rowan is taught with the goal of performing it for at least 10 hours before the surgery, it is conducted the training program after the surgery.
  Interventions: Procedure: intervention group

INTERVENTIONS:
Procedure: control group — The entire process is carried out according to Severance Hospital surgical protocols. The patients of control group will receive education from the research team about the importance of nutrition and exercise before and after surgery.
  Arms: control group
Procedure: intervention group — For the intervention group, the entire process is carried out according to the Severance Hospital surgical protocol, and the research team provides education before surgery on the importance of nutrition and exercise before and after surgery. In addition, the cognitive training program developed by Rowan is taught with the goal of performing it for at least 10 hours before the surgery, it is conducted the training program after the surgery.
  Arms: intervention group

SUMMARY:
This study is a prospective, single-center, randomized controlled trial to compare whether applying cognitive intervention therapy before and after surgery in elderly patients aged 65 years or older undergoing non-cardiac surgery can reduce the incidence of postoperative delirium compared to conservative treatment.

ELIGIBILITY:
Inclusion Criteria:

* Elderly patients aged 65 and above.
* Patients undergoing orthopedic, thoracic, or hepatopancreatobiliary surgery under general anesthesia with an expected surgery duration of 2 hours or more.
* Patients scheduled for arterial catheterization.

Exclusion Criteria:

* Patients with uncontrolled systemic conditions such as diabetes and hypertension.
* Those with visual impairment.
* Patients with cognitive impairment based on the MMSE-DS criteria.
* Individuals experiencing difficulty in communication.
* Those diagnosed with neurological disorders (such as brain hemorrhage, stroke, brain tumor, dementia, Parkinson's disease, cognitive impairment, depression, etc.).
* Patients diagnosed with alcohol or substance addiction.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
incidence of postoperative delirium | from postoperative day 0 to postoperative day 7
  Confusion assessment methods(CAM) will be used to assess postoperative delirium at least two times a day during the hospitalization period. Patients diagnosed with delirium using the CAM were evaluated for the duration, symptoms, and type of delirium (e.g., reduced awareness of the environment; poor cognitive skills; behavioral changes, including hallucinations, restlessness, calling out, slowed movement, or lethargy; and emotional disturbances, such as anxiety, irritability, euphoria, apathy, unpredictable mood shift, and personality changes).

SECONDARY OUTCOMES:
comprehensive geriatric assessment(CGA), | from postoperative day 0 to postoperative day 7
  Core component of CGA are as follows : functional capacity, fall risk, cognition, mood, polypharmacy, social support, financial concerns, goals of care, and advance care preferences.
duration of delirium | from postoperative day 0 to postoperative day 7
type of delirium | from postoperative day 0 to postoperative day 7
total score of QOR-40 | from postoperative day 0 to postoperative day 7
  The Quality of Recovery-40 (QoR-40) is a commonly utilized self-assessment questionnaire designed for postoperative patients. This survey is self-administered and aims to gather feedback from individuals about the quality of their recovery in the postoperative phase.
  The QoR-40 is divided into categories such as emotional status, physical comfort, psychological support, physical independence, and pain. Max score of QoR-40 is 200.

CONTACTS AND LOCATIONS:
Overall Officials: Bon-Nyeo Koo, Principal Investigator — Department of Anesthesiology and Pain Medicine Yonsei University College of Medicine
Locations (1):
- Department of Anesthesiology and Pain Medicine Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No